CLINICAL TRIAL: NCT02709382
Title: A Single-dose Study to Investigate the Pharmacokinetics of Intravenous FEP-TAZ in Patients With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: Clinartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: W-4282-104
Record Dates: First submitted 2016-02-26; First posted 2016-03-16 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Cefepime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FEP-TAZ (Experimental): Cefepime and Tazobactam combination; IV infusion over a period of 90 minutes Healthy subjects, Mild and Moderate RI: 4 g (2 g FEP and 2 g TAZ) Severe RI and patients on HD: 2 g (1 g FEP and 1 g TAZ)
  Interventions: Drug: Cefepime and Tazobactam combination

INTERVENTIONS:
Drug: Cefepime and Tazobactam combination

SUMMARY:
This is a Phase 1, open label, single-dose, pharmacokinetic study to be conducted in male and female subjects with normal and impaired renal function. The study will be composed of five groups of patients with mild (6 patients), moderate (6 patients), severe (6 patients) renal impairment, end stage renal disease patients on hemodialysis (6 patients) and their respective matched controls in 1:1 ratio (24 healthy subjects with normal renal function).

ELIGIBILITY:
Inclusion Criteria:

-Patients with renal impairment: mild, moderate, severe and patients on hemodialysis) that has been stable OR

* Healthy Subjects:
* Have normal renal function
* No evidence of any disease or condition that may affect pharmacokinetics of FEP-TAZ.

Exclusion Criteria:

* Evidence of hepatorenal or nephritic syndrome
* Any clinically significant abnormal findings on medical history, physical examination,or clinical laboratory tests (other than those associated with controlled diabetes,hypertension, hypercholesterolemia, dyslipidemia, or renal impairment or related or causative diseases)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
plasma concentrations (Cmax) | 48 hrs
Tmax The elimination half-life (t1/2), | 48 hrs

SECONDARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values | 14 days
Number of Participants With Adverse Events | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami,Division of Clinical Pharmacology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Preston RA, Mamikonyan G, Mastim M, Garg D, Kemper CJ, Xu A, Yeole R, Chavan R, Friedland HD, Bhatia A. Single-Center Investigation of the Pharmacokinetics of WCK 4282 (Cefepime-Tazobactam Combination) in Renal Impairment. Antimicrob Agents Chemother. 2019 Sep 23;63(10):e00873-19. doi: 10.1128/AAC.00873-19. Print 2019 Oct. PMID 31332068